CLINICAL TRIAL: NCT01244906
Title: A Phase II Trial of Post-Transplant Cyclophosphamide and Sirolimus for Graft-versus-host Disease (GVHD) Prophylaxis Following Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Post-transplant Cyclophosphamide and Sirolimus Following Reduced Intensity Conditioning (RIC) Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 911
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-01

CONDITIONS: Hematologic Neoplasms
Keywords: Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Myelofibrosis; Acute Lymphocytic Leukemia; Acute Lymphoblastic Lymphoma; Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Low-grade non-Hodgkin's Lymphoma; Mantle Cell Lymphoma; Hodgkin Lymphoma; Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Hodgkin Disease; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced Intensity Allogeneic Stem Cell Transplantation (Experimental): All patients will receive fludarabine, busulfan and cyclophosphamide as the conditioning regimen prior to an allo SCT. Patients will then receive 2 doses of cyclophosphamide post-transplant and utilize sirolimus and mycophenolate mofetil (in mismatched transplants) as GVHD prophylaxis.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Patients will receive fludarabine, busulfan and cyclophosphamide as the conditioning regimen prior to an allo SCT. Patients will then receive 2 doses of cyclophosphamide post-transplant and utilize sirolimus and mycophenolate mofetil (in mismatched transplants) as GVHD prophylaxis.

SUMMARY:
This trial will evaluate the safety and efficacy of post-transplant Cy and sirolimus following reduced intensity allogeneic SCT. It is hoped that the combination of a reduced intensity preparative regimen with a calcineurin-free GVHD prophylaxis regimen will decrease the risk of acute and chronic GVHD, by both limiting mucosal toxicity and augmenting immune reconstitution, thereby improving the safety of the procedure. The past experience with post-transplant Cy suggests that SCT recipients will attain rapid donor T cell chimerism, which the investigators hope will translate into improved disease control through the well documented graft-versus-malignancy effects of donor T cells.

ELIGIBILITY:
Inclusion Criteria:

* Availability of a 7/8 or 8/8 (HLA-A, B, C, DR) related or unrelated donor
* Age 18-75
* One of the following high-risk malignancies
* Chronic Myelogenous Leukemia
* Acute Myelogenous Leukemia
* Myelodysplastic Syndrome
* Myelofibrosis
* Acute Lymphocytic Leukemia
* Acute Lymphoblastic Lymphoma
* Chronic Lymphocytic Leukemia
* Prolymphocytic Leukemia
* Low-grade non-Hodgkin's Lymphoma
* Mantle Cell Lymphoma
* Hodgkin Lymphoma
* Myeloma

Exclusion Criteria:

* Poor cardiac function (EF <40%)
* Poor pulmonary function (FEV1 and FVC <50% predicted)
* Poor liver function (bilirubin >/= 2 mg/dl not due to hemolysis, Gilbert's or primary malignancy)
* Poor renal function (creatinine >/= 2 mg/dl or creatinine clearance <40mL/min)
* Karnofsky status <70%
* HIV positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Szydlo R, Goldman JM, Klein JP, Gale RP, Ash RC, Bach FH, Bradley BA, Casper JT, Flomenberg N, Gajewski JL, Gluckman E, Henslee-Downey PJ, Hows JM, Jacobsen N, Kolb HJ, Lowenberg B, Masaoka T, Rowlings PA, Sondel PM, van Bekkum DW, van Rood JJ, Vowels MR, Zhang MJ, Horowitz MM. Results of allogeneic bone marrow transplants for leukemia using donors other than HLA-identical siblings. J Clin Oncol. 1997 May;15(5):1767-77. doi: 10.1200/JCO.1997.15.5.1767. PMID 9164184
- [Background] de Witte T, Brand R, van Biezen A, Mufti G, Ruutu T, Finke J, von dem Borne P, Vitek A, Delforge M, Alessandrino P, Harlahakis N, Russell N, Martino R, Verdonck L, Kroger N, Niederwieser D; European Blood and Marrow Transplantation Group (EBMT), Chronic Leukemia Working Party (CLWP)-MDS subcommittee. Allogeneic stem cell transplantation for patients with refractory anaemia with matched related and unrelated donors: delay of the transplant is associated with inferior survival. Br J Haematol. 2009 Sep;146(6):627-36. doi: 10.1111/j.1365-2141.2009.07809.x. Epub 2009 Jul 14. PMID 19604243
- [Background] Basara N, Schulze A, Wedding U, Mohren M, Gerhardt A, Junghanss C, Peter N, Dolken G, Becker C, Heyn S, Kliem C, Lange T, Krahl R, Ponisch W, Fricke HJ, Sayer HG, Al-Ali H, Kamprad F, Niederwieser D; East German Study Group Hematology and Oncology (OSHO). Early related or unrelated haematopoietic cell transplantation results in higher overall survival and leukaemia-free survival compared with conventional chemotherapy in high-risk acute myeloid leukaemia patients in first complete remission. Leukemia. 2009 Apr;23(4):635-40. doi: 10.1038/leu.2008.352. Epub 2009 Jan 8. PMID 19151786
- [Background] Mielcarek M, Storer BE, Sandmaier BM, Sorror ML, Maloney DG, Petersdorf E, Martin PJ, Storb R. Comparable outcomes after nonmyeloablative hematopoietic cell transplantation with unrelated and related donors. Biol Blood Marrow Transplant. 2007 Dec;13(12):1499-507. doi: 10.1016/j.bbmt.2007.09.004. PMID 18022580
- [Background] Taylor PA, Lees CJ, Blazar BR. The infusion of ex vivo activated and expanded CD4(+)CD25(+) immune regulatory cells inhibits graft-versus-host disease lethality. Blood. 2002 May 15;99(10):3493-9. doi: 10.1182/blood.v99.10.3493. PMID 11986199
- [Background] Edinger M, Hoffmann P, Ermann J, Drago K, Fathman CG, Strober S, Negrin RS. CD4+CD25+ regulatory T cells preserve graft-versus-tumor activity while inhibiting graft-versus-host disease after bone marrow transplantation. Nat Med. 2003 Sep;9(9):1144-50. doi: 10.1038/nm915. Epub 2003 Aug 17. PMID 12925844
- [Background] Trenado A, Charlotte F, Fisson S, Yagello M, Klatzmann D, Salomon BL, Cohen JL. Recipient-type specific CD4+CD25+ regulatory T cells favor immune reconstitution and control graft-versus-host disease while maintaining graft-versus-leukemia. J Clin Invest. 2003 Dec;112(11):1688-96. doi: 10.1172/JCI17702. PMID 14660744
- [Background] Zhao D, Zhang C, Yi T, Lin CL, Todorov I, Kandeel F, Forman S, Zeng D. In vivo-activated CD103+CD4+ regulatory T cells ameliorate ongoing chronic graft-versus-host disease. Blood. 2008 Sep 1;112(5):2129-38. doi: 10.1182/blood-2008-02-140277. Epub 2008 Jun 12. PMID 18550852
- [Background] Zorn E, Kim HT, Lee SJ, Floyd BH, Litsa D, Arumugarajah S, Bellucci R, Alyea EP, Antin JH, Soiffer RJ, Ritz J. Reduced frequency of FOXP3+ CD4+CD25+ regulatory T cells in patients with chronic graft-versus-host disease. Blood. 2005 Oct 15;106(8):2903-11. doi: 10.1182/blood-2005-03-1257. Epub 2005 Jun 21. PMID 15972448
- [Background] Rieger K, Loddenkemper C, Maul J, Fietz T, Wolff D, Terpe H, Steiner B, Berg E, Miehlke S, Bornhauser M, Schneider T, Zeitz M, Stein H, Thiel E, Duchmann R, Uharek L. Mucosal FOXP3+ regulatory T cells are numerically deficient in acute and chronic GvHD. Blood. 2006 Feb 15;107(4):1717-23. doi: 10.1182/blood-2005-06-2529. Epub 2005 Nov 8. PMID 16278306
- [Background] Rezvani K, Mielke S, Ahmadzadeh M, Kilical Y, Savani BN, Zeilah J, Keyvanfar K, Montero A, Hensel N, Kurlander R, Barrett AJ. High donor FOXP3-positive regulatory T-cell (Treg) content is associated with a low risk of GVHD following HLA-matched allogeneic SCT. Blood. 2006 Aug 15;108(4):1291-7. doi: 10.1182/blood-2006-02-003996. Epub 2006 Apr 20. PMID 16627754
- [Background] Coenen JJ, Koenen HJ, van Rijssen E, Kasran A, Boon L, Hilbrands LB, Joosten I. Rapamycin, not cyclosporine, permits thymic generation and peripheral preservation of CD4+ CD25+ FoxP3+ T cells. Bone Marrow Transplant. 2007 May;39(9):537-45. doi: 10.1038/sj.bmt.1705628. Epub 2007 Mar 12. PMID 17351648
- [Background] Zeiser R, Nguyen VH, Beilhack A, Buess M, Schulz S, Baker J, Contag CH, Negrin RS. Inhibition of CD4+CD25+ regulatory T-cell function by calcineurin-dependent interleukin-2 production. Blood. 2006 Jul 1;108(1):390-9. doi: 10.1182/blood-2006-01-0329. Epub 2006 Mar 7. PMID 16522809
- [Background] Lehnert S, Rybka WB. Amplification of the graft-versus-host reaction by cyclophosphamide: dependence on timing of drug administration. Bone Marrow Transplant. 1994 Apr;13(4):473-7. PMID 8019473
- [Background] Mayumi H. [Cyclophosphamide-induced immunological tolerance: an overview]. Nihon Geka Gakkai Zasshi. 1996 Dec;97(12):1097-108. Japanese. PMID 9032788
- [Background] Mayumi H, Himeno K, Tanaka K, Tokuda N, Fan JL, Nomoto K. Drug-induced tolerance to allografts in mice. XII. The relationships between tolerance, chimerism, and graft-versus-host disease. Transplantation. 1987 Aug;44(2):286-90. doi: 10.1097/00007890-198708000-00021. PMID 3307052
- [Background] Luznik L, Jalla S, Engstrom LW, Iannone R, Fuchs EJ. Durable engraftment of major histocompatibility complex-incompatible cells after nonmyeloablative conditioning with fludarabine, low-dose total body irradiation, and posttransplantation cyclophosphamide. Blood. 2001 Dec 1;98(12):3456-64. doi: 10.1182/blood.v98.12.3456. PMID 11719388
- [Background] Luznik L, Engstrom LW, Iannone R, Fuchs EJ. Posttransplantation cyclophosphamide facilitates engraftment of major histocompatibility complex-identical allogeneic marrow in mice conditioned with low-dose total body irradiation. Biol Blood Marrow Transplant. 2002;8(3):131-8. doi: 10.1053/bbmt.2002.v8.pm11939602.
- [Background] O'Donnell PV, Luznik L, Jones RJ, Vogelsang GB, Leffell MS, Phelps M, Rhubart P, Cowan K, Piantados S, Fuchs EJ. Nonmyeloablative bone marrow transplantation from partially HLA-mismatched related donors using posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2002;8(7):377-86. doi: 10.1053/bbmt.2002.v8.pm12171484.
- [Background] Luznik L, Bolanos-Meade J, Zahurak M, Chen AR, Smith BD, Brodsky R, Huff CA, Borrello I, Matsui W, Powell JD, Kasamon Y, Goodman SN, Hess A, Levitsky HI, Ambinder RF, Jones RJ, Fuchs EJ. High-dose cyclophosphamide as single-agent, short-course prophylaxis of graft-versus-host disease. Blood. 2010 Apr 22;115(16):3224-30. doi: 10.1182/blood-2009-11-251595. Epub 2010 Feb 2. PMID 20124511
- [Background] Uberti JP, Ayash L, Braun T, Reynolds C, Silver S, Ratanatharathorn V. Tacrolimus as monotherapy or combined with minidose methotrexate for graft-versus-host disease prophylaxis after allogeneic peripheral blood stem cell transplantation: long-term outcomes. Bone Marrow Transplant. 2004 Sep;34(5):425-31. doi: 10.1038/sj.bmt.1704594. PMID 15273705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Started | 26
Completed | 18
Not Completed | 8
Not completed — Death | 2
Not completed — Progression of disease post treatment | 6

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 73]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Incidence of GVHD
Description: To estimate the incidence of graft-versus-host disease (GVHD) when utilizing post-transplant cyclophosphamide (Cy) and sirolimus for GVHD prophylaxis following reduced intensity allogeneic hematopoietic stem cell transplantation (SCT) in patients with high risk hematologic malignancies.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
participants | 12

2. Secondary Outcome: Incidence of Absolute Neutrophil Count (ANC)/Platelet Engraftment
Description: To estimate the incidence of neutrophil and platelet engraftment
Time Frame: Approximately Day 30
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
participants | 26

3. Secondary Outcome: Number of Participants With Non-Relapse Mortality
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
participants | 1

4. Secondary Outcome: Number of Patients With Disease Free Survival at 2 Years
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
participants | 17

5. Secondary Outcome: Number of Patients to Achieve Full Donor Chimerism
Description: Characterize rate of achievement of full donor chimerism
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
participants | 26

6. Secondary Outcome: Number of Patients With Overall Survival at 2 Years.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 26
participants | 19

ADVERSE EVENTS:
Arm/Group | Reduced Intensity Allogeneic Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Intensity Allogeneic Stem Cell Transplantation (N=26)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute Cholecystitis (Gastrointestinal disorders) | 1 (1)
GI bleeding (Gastrointestinal disorders) | 2 (2)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cellulitis (Vascular disorders) | 1 (1)
VOD (Hepatobiliary disorders) | 1 (1)
Severe Hyperglycemia (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced Intensity Allogeneic Stem Cell Transplantation (N=26)
Nausea (Gastrointestinal disorders) | 24
"cold sweats" (General disorders) | 2
"cold" feeling (General disorders) | 2
abdominal bloating (Gastrointestinal disorders) | 8
abdominal cramps (Gastrointestinal disorders) | 8
abdominal discomfort/pain (Gastrointestinal disorders) | 14
abdominal distention (Gastrointestinal disorders) | 13
abdominal tenderness (Gastrointestinal disorders) | 5
agitation (Psychiatric disorders) | 3
increased alkaline phosphatase (Hepatobiliary disorders) | 17
alopecia (General disorders) | 3
increased alanine aminotransferase (Hepatobiliary disorders) | 18
neutropenia (Blood and lymphatic system disorders) | 26
anemia (Blood and lymphatic system disorders) | 26
anorexia/decreased oral intake (Gastrointestinal disorders) | 11
anxiety (Psychiatric disorders) | 21
arm pain (Musculoskeletal and connective tissue disorders) | 3
ascites (Gastrointestinal disorders) | 5
increased aspartate aminotransferase (Hepatobiliary disorders) | 14
ataxia (Musculoskeletal and connective tissue disorders) | 11
back pain (Musculoskeletal and connective tissue disorders) | 12
bacteremia (Infections and infestations) | 6
bilateral knee pain (Musculoskeletal and connective tissue disorders) | 2
BKV cystitis (Infections and infestations) | 12
bladder cramping (Renal and urinary disorders) | 2
bladder pain (Renal and urinary disorders) | 7
bladder spasms (Renal and urinary disorders) | 6
bloody stool (Gastrointestinal disorders) | 2
blurry vision (Eye disorders) | 4
benign prostatic hyperplasia (Renal and urinary disorders) | 2
bradycardia (Cardiac disorders) | 6
bruising (Skin and subcutaneous tissue disorders) | 10
clostridium difficile colitis (Gastrointestinal disorders) | 4
cellulitis (Infections and infestations) | 3
chest pressure (Cardiac disorders) | 2
chills/rigors (General disorders) | 14
CMV reactivation (Infections and infestations) | 2
confusion (Psychiatric disorders) | 2
constipation (Gastrointestinal disorders) | 13
dry cough (Respiratory, thoracic and mediastinal disorders) | 17
coarse breath sounds (Respiratory, thoracic and mediastinal disorders) | 3
increased creatinine (Renal and urinary disorders) | 9
central venous catheter pain (General disorders) | 15
central venous catheter site drainage (General disorders) | 5
central venous catheter site erythema (General disorders) | 8
deconditioning (General disorders) | 10
decreased appetite (Metabolism and nutrition disorders) | 18
decreased bowel movement frequency (Gastrointestinal disorders) | 2
decreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 10
decreased fluid intake (Metabolism and nutrition disorders) | 5
depression (Psychiatric disorders) | 13
diaphoretic skin (Skin and subcutaneous tissue disorders) | 2
diarrhea (Gastrointestinal disorders) | 23
dysphagia (Gastrointestinal disorders) | 7
dizziness (Nervous system disorders) | 9
drowsiness (Nervous system disorders) | 12
dry eyes (Eye disorders) | 6
dry lips (Gastrointestinal disorders) | 2
dry mouth (Gastrointestinal disorders) | 9
dry skin (Skin and subcutaneous tissue disorders) | 10
deep venous thrombosis (Vascular disorders) | 2
dysuria (Renal and urinary disorders) | 16
ear fullness/pressure (Ear and labyrinth disorders) | 2
electrolyte wasting syndrome (Metabolism and nutrition disorders) | 2
enlarged lymph nodes (Blood and lymphatic system disorders) | 2
epigastric pain (Gastrointestinal disorders) | 2
epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
esophagitis (Gastrointestinal disorders) | 2
excoriation (Skin and subcutaneous tissue disorders) | 3
facial edema (General disorders) | 2
fatigue (General disorders) | 22
fever (General disorders) | 20
flat affect (Psychiatric disorders) | 7
fluid overload (Vascular disorders) | 9
facial flushing (Vascular disorders) | 4
folliculitis (Skin and subcutaneous tissue disorders) | 4
gas/flatulence (Gastrointestinal disorders) | 3
generalized achiness (Musculoskeletal and connective tissue disorders) | 7
generalized skin erythema (Skin and subcutaneous tissue disorders) | 4
GERD (Gastrointestinal disorders) | 19
skin GVHD (Immune system disorders) | 11
gut GVHD (Immune system disorders) | 2
hallucinations (Psychiatric disorders) | 2
headache (Nervous system disorders) | 16
hematoma (Vascular disorders) | 2
hematuria (Renal and urinary disorders) | 12
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
perirectal bleeding/hemorrhage (Gastrointestinal disorders) | 7
hemorrhodial edema (Gastrointestinal disorders) | 2
hemorrhodial pain (Gastrointestinal disorders) | 4
hemorrhoids (Gastrointestinal disorders) | 7
hernia (Musculoskeletal and connective tissue disorders) | 2
hives (Skin and subcutaneous tissue disorders) | 2
hyperactive bowel sounds (Gastrointestinal disorders) | 6
hyperbilirubinemia (Hepatobiliary disorders) | 11
hypercalcemia (Metabolism and nutrition disorders) | 4
hyperglycemia (Metabolism and nutrition disorders) | 26
hyperkalemia (Metabolism and nutrition disorders) | 3
hypernatremia (Metabolism and nutrition disorders) | 14
hyperpigmentation (Skin and subcutaneous tissue disorders) | 7
hypertension (Cardiac disorders) | 16
hypoalbuminemia (Metabolism and nutrition disorders) | 20
hypocalcemia (Metabolism and nutrition disorders) | 20
hypoglycemia (Metabolism and nutrition disorders) | 2
hypokalemia (Metabolism and nutrition disorders) | 18
hypomagnesemia (Metabolism and nutrition disorders) | 16
hyponatremia (Metabolism and nutrition disorders) | 9
hypotension (Cardiac disorders) | 13
hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
stool incontinence (Gastrointestinal disorders) | 4
increased respiration rate (Respiratory, thoracic and mediastinal disorders) | 2
insomnia (Psychiatric disorders) | 13
joint aches (Musculoskeletal and connective tissue disorders) | 3
lower-extremity edema (General disorders) | 17
leg pain (Musculoskeletal and connective tissue disorders) | 2
lethargy (Nervous system disorders) | 10
limited mobility (Musculoskeletal and connective tissue disorders) | 5
lip edema (General disorders) | 2
loss of coordination/balance (Nervous system disorders) | 5
lung crackles (Respiratory, thoracic and mediastinal disorders) | 10
lymphadenopathy (Blood and lymphatic system disorders) | 2
malnutrition (Gastrointestinal disorders) | 2
metabolic acidosis (Metabolism and nutrition disorders) | 2
mouth sores (Gastrointestinal disorders) | 9
mouth tenderness (Gastrointestinal disorders) | 10
MRSE bacteremia (Infections and infestations) | 3
mucositis (Gastrointestinal disorders) | 15
muscle weakness (Musculoskeletal and connective tissue disorders) | 2
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10
nasal drainage (Respiratory, thoracic and mediastinal disorders) | 7
neuropathy (Nervous system disorders) | 7
febrile neutropenia (Blood and lymphatic system disorders) | 15
nocturia (Renal and urinary disorders) | 2
oral erythema (Skin and subcutaneous tissue disorders) | 3
oral thrush (Vascular disorders) | 2
orthostatic hypotension (Cardiac disorders) | 2
pain during defication (Gastrointestinal disorders) | 2
pain with breathing (Respiratory, thoracic and mediastinal disorders) | 3
hip pain (Musculoskeletal and connective tissue disorders) | 2
foot pain (Musculoskeletal and connective tissue disorders) | 2
lower-extremity pain (Musculoskeletal and connective tissue disorders) | 2
neck pain (Musculoskeletal and connective tissue disorders) | 2
pelvic pain (Musculoskeletal and connective tissue disorders) | 3
shoulder pain (Musculoskeletal and connective tissue disorders) | 4
throat pain (Gastrointestinal disorders) | 13
pale skin (Skin and subcutaneous tissue disorders) | 3
parainfluenza (Respiratory, thoracic and mediastinal disorders) | 3
penile lesions (Skin and subcutaneous tissue disorders) | 3
perihepatic ascites (Hepatobiliary disorders) | 2
periorbital edema (Eye disorders) | 2
periorbital redness (Eye disorders) | 2
peripheral edema (General disorders) | 3
perirectal irritation (Gastrointestinal disorders) | 4
perirectal pain (Gastrointestinal disorders) | 4
petechiae (Blood and lymphatic system disorders) | 2
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
pleuritic chest pain (Cardiac disorders) | 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 5
post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 4
pruritus (Skin and subcutaneous tissue disorders) | 17
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5
pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 2
pulmonary opacites (Respiratory, thoracic and mediastinal disorders) | 4
rash (Skin and subcutaneous tissue disorders) | 20
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 5
restless leg syndrome (Nervous system disorders) | 2
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6
rhinovirus/URI (Respiratory, thoracic and mediastinal disorders) | 7
rhonchi (Respiratory, thoracic and mediastinal disorders) | 5
ribcage tenderness (Musculoskeletal and connective tissue disorders) | 2
seasonal allergies (General disorders) | 9
sedation (Nervous system disorders) | 4
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7
sinus drainage (Respiratory, thoracic and mediastinal disorders) | 14
sinus pressure (Respiratory, thoracic and mediastinal disorders) | 3
chronic sinusitis (Respiratory, thoracic and mediastinal disorders) | 4
skin abrasion (Skin and subcutaneous tissue disorders) | 3
skin color changes (Skin and subcutaneous tissue disorders) | 3
skin erythema (Skin and subcutaneous tissue disorders) | 3
skin lesions (Skin and subcutaneous tissue disorders) | 4
skin sensitivity (Skin and subcutaneous tissue disorders) | 2
skin tear (Skin and subcutaneous tissue disorders) | 2
skin tenderness (Skin and subcutaneous tissue disorders) | 2
sneezing (Respiratory, thoracic and mediastinal disorders) | 2
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 15
splenomegaly (General disorders) | 2
staphylococcus epidermis bacteremia (Infections and infestations) | 2
steroid-induced diabetes (Metabolism and nutrition disorders) | 6
stomatitis (Gastrointestinal disorders) | 3
suprapubic tenderness (Musculoskeletal and connective tissue disorders) | 2
sweats (Nervous system disorders) | 6
tachycardia (Cardiac disorders) | 17
taste changes (General disorders) | 7
thrombocytopenia (Blood and lymphatic system disorders) | 26
tremors (Nervous system disorders) | 5
unsteady gait (Nervous system disorders) | 2
urinary frequency (Renal and urinary disorders) | 15
urinary hesitancy (Renal and urinary disorders) | 3
urinary incontinence (Renal and urinary disorders) | 4
urinary retention (Renal and urinary disorders) | 5
urinary urgency (Renal and urinary disorders) | 6
urinary tract infection (Renal and urinary disorders) | 2
visual changes (Nervous system disorders) | 4
veno-occlusive disease (Hepatobiliary disorders) | 2
volume depletion (General disorders) | 3
vomiting (Gastrointestinal disorders) | 21
VRE positive (Infections and infestations) | 6
leukopenia (Blood and lymphatic system disorders) | 26
generalized weakness (General disorders) | 15
weight gain (Investigations) | 5
weight loss (Investigations) | 12
wheezing (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes